CLINICAL TRIAL: NCT01215461
Title: Evaluation of Factors Associated With Mortality in Neonates
Brief Title: Factors Associated With Mortality in Neonates
Status: Completed | Type: Observational
Sponsor: Pediatrix (Other)
Responsible Party: Sponsor
Other Study IDs: PDX-001-10
Record Dates: First submitted 2010-10-05; First posted 2010-10-06 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Neonatal Mortality
Keywords: Neonatal mortality; Preterm birth; Low gestational age; VLBW
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to better understand the factors associated with mortality and identify potentially preventable causes of death in neonates who die after receiving health care. As a result, an improved neonatal mortality classification system may be defined.

ELIGIBILITY:
Inclusion Criteria:

* Neonates for whom healthcare was provided
* Born alive
* Neonate greater than or equal to 22 0/7 weeks estimated gestational age

Exclusion Criteria:

* Stillborn
* Fetal demise
* Neonates less than or equal to 21 6/7 weeks estimated gestational age

Ages: 22 Weeks to 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates for whom healthcare was provided.
Sampling Method: Non-Probability Sample
Enrollment: 645 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To better understand the factors associated with mortality and identify potentially preventable causes of death in neonates who die after receiving health care. | neonatal outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Providence Alaska Medical Center, Anchorage, Alaska, United States